CLINICAL TRIAL: NCT00412555
Title: An Open-label Multi-center Trial of Oseltamivir for the Seasonal Prophylaxis of Influenza in Children.
Brief Title: A Study of Tamiflu (Oseltamivir) for Seasonal Prophylaxis of Influenza in Children.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NV20236
Record Dates: First submitted 2006-12-15; First posted 2006-12-18 (Estimated); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: oseltamivir [Tamiflu]

INTERVENTIONS:
Drug: oseltamivir [Tamiflu] — 30-75mg po daily for 6 weeks

SUMMARY:
This study will evaluate the safety of Tamiflu, when used for the prevention of influenza in children during the flu season. Children who would benefit from influenza prophylaxis when influenza is circulating in the community will receive treatment with Tamiflu syrup (or capsules) 30mg-75mg once daily (dependent on body weight) for 6 weeks. Safety data and influenza symptoms will be recorded throughout the study. The anticipated time on study treatment is <3 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* males or females, 1-12 years of age;
* candidate for seasonal prophylaxis;
* negative rapid diagnostic test for influenza at baseline.

Exclusion Criteria:

* symptoms suggestive of influenza-like illness;
* positive rapid diagnostic test for influenza;
* antiviral treatment for influenza in 2 weeks prior to randomization.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2006-12; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
AEs, laboratory parameters, vital signs. | Throughout study
Percentage of patients with laboratory confirmed clinical influenza | Throughout study

SECONDARY OUTCOMES:
Percentage of subjects with asymptomatic influenza; percentage with an influenza-like illness. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- United States (4):
  - West Palm Beach, Florida
  - Pittsburgh, Pennsylvania
  - Jackson, Tennessee
  - El Paso, Texas
- Coquitlam, British Columbia, Canada
- Aalborg, Denmark

REFERENCES:
- [Derived] Reisinger K, Shu D, Cupelli L, Marcadis I, Dutkowski R. Safety and tolerability of a 6-week course of oseltamivir prophylaxis for seasonal influenza in children. Influenza Other Respir Viruses. 2013 Jan;7(1):11-3. doi: 10.1111/j.1750-2659.2012.00367.x. Epub 2012 Apr 23. PMID 22520945